CLINICAL TRIAL: NCT07257042
Title: The Clinical Investigation of a Toothpaste Containing 8% Arginine Compared to Colgate Cavity Protection Toothpaste in Reducing Dentinal Hypersensitivity - an Eight-week Clinical Study in the US
Brief Title: Oothpaste Containing 8% Arginine Compared to Colgate Cavity Protection Toothpaste in Reducing Dentinal Hypersensitivity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO-2025-06-SEN-TOM-ARG-YPZ
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Hypersensitivity
MeSH Terms: conditions — Hypersensitivity | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Test 1 toothpaste (Experimental): subjects will brush with assigned toothpaste morning & night
  Interventions: Drug: Toothpaste containing 8% Arginine
- Control toothpaste (Active Comparator): subjects will brush with assigned toothpaste morning & night
  Interventions: Drug: Colgate Cavity Protection Toothpaste

INTERVENTIONS:
Drug: Toothpaste containing 8% Arginine — Brush twice daily (morning and evening) for one full minute Cover the entire length of bristles with toothpaste
  Arms: Test 1 toothpaste
Drug: Colgate Cavity Protection Toothpaste — Brush twice daily (morning and evening) for one full minute Cover the entire length of bristles with toothpaste
  Arms: Control toothpaste

SUMMARY:
The objective of this study is to assess clinical efficacy of a toothpaste containing 8% arginine (Colgate-Palmolive Company, New York, NY, USA) to provide dental hypersensitivity relief (tactile and air blast) in comparison to Colgate Cavity Protection Toothpaste (Colgate-Palmolive Company, New York, NY, USA) over an eight-week period.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, ages 18-70, inclusive.
* Availability for the eight-week duration of the study.
* Two sensitive teeth, which must be anterior to the molars, and demonstrate cervical erosion/abrasion or gingival recession.
* Qualifying response to tactile stimuli (Yeaple probe) as defined by a score between 10-50 gms. of force.
* Qualifying response to the air blast stimuli as defined by a score of 2 or 3 on the Schiff Cold Air Sensitivity Scale.
* Subjects need to satisfy the qualifying response to stimuli for both the parameters assessed (tactile or air) on two teeth to be entered into the study.
* Good general health with no known allergies to products being tested.
* Use of a non-desensitizing dentifrice for three months prior to entry into the study.
* Signed Informed Consent Form

Exclusion Criteria:

* Gross oral pathology, chronic disease, or history of allergy to test products.
* Advanced periodontal disease or treatment for periodontal disease (including surgery) within the past twelve months.
* Sensitive teeth with a mobility greater than one.
* Teeth with extensive/defective restorations (including prosthetic crowns), suspected pulpitis, caries, cracked enamel, or used as abutments for removable partial dentures.
* Current use of anticonvulsants, antihistamines, antidepressants, sedatives, tranquilizers, anti-inflammatory drugs, or daily use of analgesics.
* Participation in a desensitizing dentifrice study or regular use of a desensitizing dentifrice within the past three months.
* Current participation in any other clinical study.
* Pregnant or lactating subjects.
* Allergies to oral care products, personal care consumer products, or their ingredients.
* Medical condition which prohibits not eating/drinking for 4 hours.
* Use in the past of the two test dentifrices.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-07-14 (Actual); Primary Completion 2025-11-04 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Tactile stimulation with a Yeaple Probe. treatment Tactile and Air Blast Hypersensitivity scores. The mean Tactile and Air Blast Hypersensitivity will be computed and summarized | Baseline 4 week & 8 week
  Sensitivity will be defined by a score in the range of 10-50 gms. of force
Schiff Cold Air Sensitivity Scale | Baseline 4 week & 8 week
  Sensitivity will be defined by a score of 2 or 3 on the Schiff Cold Air Sensitivity Scale

CONTACTS AND LOCATIONS:
Overall Officials: Yiming LI, DDS, PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No